CLINICAL TRIAL: NCT06462599
Title: Association of Osteopontin Gene Polymorphisms With Susceptibility and Prognosis of Ischemic Stroke in Egyptian Patients
Brief Title: Osteopontin Gene Polymorphism in Stroke Patients in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madonna Nabil, Assistant lecturer, Assiut University
Other Study IDs: Gene polymorphisms in stroke
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from stroke patients within 24 hrs of stroke and normal volunteers.
  Two samples will be collected serum and plasma; five ml whole blood from patients and normal volunteers and centrifuge serum samples at 1500 rpm 10 min then will be stored at - 80 °C until the day of the analysis.
  Plasma samples will be stored at - 80 °C until the day of the analysis without centrifugation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with ischaemic stroke
  Interventions: Genetic: Gene polymorphism from blood samples
- Control: Healthy individuals
  Interventions: Genetic: Gene polymorphism from blood samples

INTERVENTIONS:
Genetic: Gene polymorphism from blood samples — Blood samples will be collected from stroke patients within 24 hrs of stroke and normal volunteers.
  Two samples will be collected serum and plasma; five ml whole blood from patients and normal volunteers and centrifuge serum samples at 1500 rpm 10 min then will be stored at - 80 °C until the day of the analysis.
  Plasma samples will be stored at - 80 °C until the day of the analysis without centrifugation

SUMMARY:
This study aims to investigate the correlation of serum osteopontin level as a predictior and a prognostic factor in upper egyptian patients and correlation between Osteopontin Gene Polymorphisms and serum level of osteopontin in ischaemic stroke patients

DETAILED DESCRIPTION:
The Global Burden of Disease estimated that one person in four aged 25 years will have a stroke in the rest of her/his life. Among them, ischemic stroke (IS) represents 80%.

Stroke is accompanied by a neuroinflammatory response involving immune system. These long-term processes following IS are still far from being understood. So, despite the significant improvement in the diagnosis and treatment of IS, the disability and mortality rate of IS are still rising. An assessment of the prognostic risk of IS should be carried out as early as possible and corresponding interventions should be adopted clinically, in order to have a significant impact on the prognosis of patients with IS.

Predicting the outcome in individual patients solely based on clinical and radiological parameters is challenging for clinicians. Measuring blood biomarkers associated with inflammation, endothelial function, matrix remodeling, and immune functions, may improve prediction performance .

Osteopontin (OPN) is a matricellular protein participating in many physiological and pathologic processes including wound healing, bone turnover, tumor genesis, inflammation, and immune responses . It is well accepted that OPN is an important mediator in stroke pathophysiology. OPN expression is upregulated in microglia surrounding the infarcted area and in microglia and infiltrating macrophages in the infarct area. OPN and microglia seems to exhibit an intimate relationship in stroke with rather beneficial functions for the clinical outcome. However, the role of OPN in stroke-related diseases as atherosclerosis and diabetes should be further disentangled as in this early phase of disease OPN may ultimately culminate in cerebrovascular dysfunction. OPN may exert opposing effects and should be therefore addressed differently.

ELIGIBILITY:
Inclusion Criteria:

* For acute ischemic stroke cases:

( Acute ischemic stroke will be defined as an episode of focal neurological deficits lasting for more than 24 hour with relevant lesion in brain computerized tomography (CT) or magnetic resonance (MR) image>)

1- both sex 2- Age between 18 to 70 years old. 3-symptoms suggestive of acute ischemic stroke: presenting within 24 hours of onset of these symptoms

* For old ischemic stroke:

  1. both sex
  2. Age between 18 to 70 years old.
  3. Duration of3to 6 month of development of ischemic symptoms
* For control cases:

  1. both sex
  2. Healthy people
  3. Age: above 18 years old

     Exclusion Criteria:

     Patients with a previous history of stroke; Patients with hemorrhagic stroke. Patients with coronary heart disease, heart failure, chronic inflammation, intracranial infection/brain tumor and malignant tumor.

     Patients with liver, kidney and other important organ dysfunction. Patients with severe abnormal coagulation function

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: we will enrol 72 participants; 36 stroke patients and 36 control cases (age matched) recruited among the attendants of Neurology department, Assiut University Hospital, adult age.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Measure osteopontin level in ischaemic stroke patients and different gene polymorphisms related to the disease | Baseline
  investigate the correlation of serum osteopontin level as a predictior and a prognostic factor in upper egyptian patients.
  Correlation between Osteopontin Gene Polymorphisms and serum level of osteopontin in ischaemic stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Michel Effat, Lecturer, Study Director — Researcher

REFERENCES:
- [Background] Jing M, Li B, Hou X, Shoba J, Li C, Liang H, Zhang X, Liu E, Yang B, Meng X. OPN gene polymorphism and the serum OPN levels confer the susceptibility and prognosis of ischemic stroke in Chinese patients. Cell Physiol Biochem. 2013;32(6):1798-807. doi: 10.1159/000356613. Epub 2013 Dec 13. PMID 24355932
- [Background] Meseguer E, Diallo D, Labreuche J, Charles H, Delbosc S, Mangin G, Monteiro Tavares L, Caligiuri G, Nicoletti A, Amarenco P. Osteopontin Predicts Three-Month Outcome in Stroke Patients Treated by Reperfusion Therapies. J Clin Med. 2020 Dec 13;9(12):4028. doi: 10.3390/jcm9124028. PMID 33322093
- [Background] Zhang Y, Wang JR, Zhang EN, Zhao ZJ. Analysis of the effect of changes in serum osteopontin levels on patients with acute cerebral infarction. Pak J Med Sci. 2024 Mar-Apr;40(4):718-722. doi: 10.12669/pjms.40.4.7045. PMID 38544995